CLINICAL TRIAL: NCT02520050
Title: The Effect of Three Different Models of Medical Nutrition Therapy (MNT) on Diabetes Control in Overweight and Obese Patients With Type 2 Diabetes: A Randomized Comparative Study. (Nutrition Path Study)
Brief Title: The Effect of 3 Different Models of MNT on DM Control in Overweight Patients With T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Metagenics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHS#: 2014-40
Record Dates: First submitted 2015-08-04; First posted 2015-08-11 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Type 2 diabetes; Obesity; Nutrition; Medical Nutrition Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Traditional MNT (Active Comparator): Will be instructed to follow a MNT plan as recommended by the ADA through consultation with a RD.
  Interventions: Behavioral: Traditional MNT
- Structured MNT (Active Comparator): Will be instructed to follow a MNT plan as applied in the Why WAIT™ program, which includes structured dietary plan, dietary modification and use of diabetes-specific meal replacement (Ultra Glucose Control®; Metagenics Inc.) three times per day.
  Interventions: Behavioral: Structured MNT
- Structured MNT plus Weekly Support (Active Comparator): Will be instructed to follow a MNT plan as applied in the Why WAIT™ program, which includes structured dietary plan, dietary modification and use of diabetes-specific meal-replacement (Ultra Glucose Control®; Metagenics Inc.) three times per day plus weekly coaching.
  Interventions: Behavioral: Structured MNT plus Weekly Support

INTERVENTIONS:
Behavioral: Traditional MNT — Will follow the nutritional recommendations set by the American Diabetes Association in 2013.
  Arms: Traditional MNT
Behavioral: Structured MNT — Will follow a meal plan developed at Joslin plus use of use of diabetes-specific nutritional formula.
  Other Names: Medical Nutritional Therapy Plan
  Arms: Structured MNT
Behavioral: Structured MNT plus Weekly Support — Will follow a meal plan developed at Joslin plus use of use of diabetes-specific nutritional formula; in addition to receiving weekly coaching from a registered dietitian
  Arms: Structured MNT plus Weekly Support

SUMMARY:
The American Diabetes Association (ADA), among other medical societies, is strongly recommending medical nutrition therapy (MNT) for prevention and management of type 2 diabetes. However, the ADA recognized that there is no "one size fits all" diet and thus recommends that MNT should be conducted through a consultation with registered dietitians (RD). Previous studies have shown that using diabetes-specific nutritional formulas, as an integral part of the MNT, lowers postprandial blood glucose levels. Through our experience from the Joslin's Weight Achievement and Intensive Treatment (Why WAIT™) program, applying MNT within a structured dietary intervention protocol has the best impact on blood glucose values and body weight. Meanwhile, the frequent use of health coaching during dietary intervention proved to be effective in managing diabetes and inducing weight loss. However, no study compared those three intervention methods in a randomized clinical study.

The aim of this study is to evaluate the effect of different models of conducting medical nutrition therapy on the glycemic control in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board/Independent Ethics Committee, and provided Health Insurance Portability and Accountability Act authorization (HIPAA) or other privacy authorization prior to any participation in study.
2. Subject states that he/she had type 2 diabetes, as evidenced by use of anti-hyperglycemic medication or managed on lifestyle intervention only with A1C >7%
3. Subject is between 30 and 80 years of age.
4. Subject on stable dose of antihyperglycemic medications for the past 3 months or lifestyle intervention
5. Subject is a male or a non-pregnant, non-lactating female, at least 6 weeks postpartum prior to screening visit. A urine pregnancy test is required for all female subjects unless she is not of childbearing potential, defined as postmenopausal for at least one year prior to screening visit or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).
6. If a female is of childbearing potential, she is practicing one of the following methods of birth control (and continued through the duration of the study):

   * Condoms, sponge, diaphragm or intrauterine device;
   * Oral or parenteral contraceptives for 3 months prior to screening visit;
   * Vasectomized partner;
   * Total abstinence from sexual intercourse.
7. Subject's BMI is > 25 kg/m2.
8. Subject has A1C between 7-10%
9. If on a chronic medication such as anti-hypertensive, lipid-lowering, thyroid medication or hormone therapy, subject has been on stable dose for at least three months prior to screening visit. These medications will not be changed during intervention unless it is mandatory.

Exclusion Criteria:

1. Subjects using exogenous insulin since insulin titration may impact the primary endpoint.
2. Subject states that he/she had a history of diabetic ketoacidosis.
3. Subject is pregnant or lactating.
4. Subject uses corticosteroid treatment with the exception of inhaled or topical steroids in the last 3 months; or antibiotics within the last 3 weeks prior to the screening visit.
5. Subject states that he/she had an active malignancy (excluding the following dermal malignancies: basal cell carcinoma, squamous cell carcinoma, carcinoma in-situ of the cervix).
6. Subject states that he/she has had a recent cardiovascular event (e.g., myocardial infarction, stroke) ≤ six months prior to screening visit; or stated history of congestive heart failure.
7. Subject states that he/she has had end stage organ failure (such as end stage renal disease) or had status post organ transplant.
8. Subject states that he/she has had a history of renal disease (Creatinine >1.5mg/dL or GFR <60 mL/min/1.73 m2).
9. Subject states that he/she has had current hepatic disease.
10. Subject has history of gastroparesis.
11. Subject states that he/she has had a chronic, contagious, infectious disease
12. Subject states that he/she has had clotting or bleeding disorders.
13. Subject is known to be allergic or intolerant to any ingredient found in the study products.
14. Subject is known to have a history of special nutritional need requiring special diet.
15. Subject is currently participating in any weight loss program.
16. Subject has used meal replacements during the 3 months prior to the start of the study.
17. Subject has history of bariatric surgery.

    -

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2015-04; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Absolute and relative change in HbA1c | 16 weeks

SECONDARY OUTCOMES:
Absolute and relative change in body weight | 16 weeks
Absolute and relative change in fasting blood glucose | 16 weeks
Absolute and relative change in lipid profile (cholesterol, HDL, LDL, triglycerides) | 16 weeks
Absolute and relative change in blood pressure | 16 weeks
Absolute and relative change in High-sensitivity C - reactive protein (hsCRP) | 16 weeks
Absolute and relative change in HOMA insulin resistance (IR) index | 16 weeks
Absolute and relative change in c-peptide level | 16 weeks
Absolute and relative change in microalbumin/creatinine ratio | 16 weeks
Absolute and relative change in fat mass | 16 weeks
Absolute and relative change in body fat percentage | 16 weeks
Absolute and relative change in waist/hip ratio | 16 weeks
Absolute and relative change in visceral fat content | 16 weeks
Absolute and relative change in dietary protein | 16 weeks
Absolute and relative change in energy intake | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Osama Hamdy, MD, PhD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mottalib A, Salsberg V, Mohd-Yusof BN, Mohamed W, Carolan P, Pober DM, Mitri J, Hamdy O. Effects of nutrition therapy on HbA1c and cardiovascular disease risk factors in overweight and obese patients with type 2 diabetes. Nutr J. 2018 Apr 7;17(1):42. doi: 10.1186/s12937-018-0351-0. PMID 29626933